CLINICAL TRIAL: NCT05827549
Title: Evaluation of Treatment Efficacy According to Risk Group in Relapsed Childhood Acute Lymphoblastic Leukemia
Acronym: ReCALL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ho Joon Im (Other)
Collaborators: Samsung Medical Center (Other); Seoul National University Hospital (Other); Severance Hospital (Other); Chonnam National University Hospital (Other); Pusan National University Yangsan Hospital (Other); Seoul St. Mary's Hospital (Other)
Responsible Party: Sponsor-Investigator, Ho Joon Im, Professor, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KPHOG_T1RALL2201
Record Dates: First submitted 2023-03-16; First posted 2023-04-25 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Acute Lymphoid Leukemia
Keywords: combination chemotherapy
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Maintenance; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Standard Risk group with B-ALL (Experimental): Reinduction -> Consolidation 1st -> Consolidation 2nd -> Repeat the Intensification course in parentheses 3 times(Intensification 1st -> Intensification 2nd -> Intensification 3rd -> Intensification 4th) -> Maintenance
  Interventions: Drug: Reinduction(4weeks); Drug: Cosolodation 1st(3weeks); Drug: Consolidation 2nd(3weeks); Drug: Intensification course; Drug: Maintenance(12 Weeks/Cycle)
- High Risk group with B-ALL (Experimental): Reinduction -> Consolidation 1st -> Consolidation 2nd -> Blinatumomab 1st -> Blinatumomab 2nd -> HSCT
  Interventions: Drug: Reinduction(4weeks); Drug: Cosolodation 1st(3weeks); Drug: Consolidation 2nd(3weeks); Drug: Blinatumomab 1st(High Risk Group)_4 Weeks; Drug: Blinatumomab 2nd (High Risk Group)_4 Weeks; Procedure: Stem Cell Transplantation
- Very high Risk with B-ALL (Experimental): Reinduction -> Blinatumomab-Salvage 1st -> Blinatumomab-Salvage 2nd -> HSCT
  Interventions: Drug: Reinduction(4weeks); Drug: Blinatumomab-Salvage 1st (Very High Risk Group)_4 Weeks; Drug: Blinatumomab-Salvage 2nd (Very High Risk Group)_4 Weeks; Drug: Intensification course
- T-ALL (Experimental): Reinduction -> Consolidation 1st -> Consolidation 2nd -> HSCT
  Interventions: Drug: Reinduction(4weeks); Drug: Cosolodation 1st(3weeks); Drug: Consolidation 2nd(3weeks); Procedure: Stem Cell Transplantation

INTERVENTIONS:
Drug: Reinduction(4weeks) — Prednisolone 60 mg/m2/day tid days 1-28, Vincristine 1.5 mg/m2 on days 1, 8, 15, 22, L-asparaginase 6,000 IU/m2(days 2-4 start, total 9 doses for 3 weeks), Idarubicin 10 mg/m2 on days 1, 8, (15~17), IT Ara-C on days 1, IT MTX on days 8, 29
Drug: Cosolodation 1st(3weeks) — Ifosfamide: 1.8 g/m2 (days 1, 2, 3, 4, 5), Etoposide: 100 mg/m2 (days 1, 2, 3, 4, 5), IT MTX on day 1
  Arms: High Risk group with B-ALL; Standard Risk group with B-ALL; T-ALL
Drug: Consolidation 2nd(3weeks) — MTX: 500 mg/m2 over 30 min followed by 1,000 mg/m2 over 23.5 hr (day 1), Ara-C: 3,000 mg/m2/dose (day 2, 3), IT MTX on day 1
  Arms: High Risk group with B-ALL; Standard Risk group with B-ALL; T-ALL
Drug: Blinatumomab 1st(High Risk Group)_4 Weeks — Blinatumomab 15 mcg/m²/day(Days: 1-28), Dexamethasone 5 mg/m2/dose on Day 1, IT MTX on day 15, 29 (CNS 1, 2 patients), TIT on day 15, 29 (CNS 3 patient)
  Arms: High Risk group with B-ALL
Drug: Blinatumomab 2nd (High Risk Group)_4 Weeks — Blinatumomab 15 mcg/m²/day(Days: 1-28), IT MTX on day 15, 29 (CNS 1, 2 patients), TIT on day 15, 29 (CNS 3 patient)
  Arms: High Risk group with B-ALL
Drug: Blinatumomab-Salvage 1st (Very High Risk Group)_4 Weeks — Blinatumomab 9 mcg/day(Weight ≥ 45kg) or 5 mcg/m²/day(Weight < 45kg) on 1-7 days, 28 mcg/day(Weight ≥ 45kg) or 15 mcg/m²/day(Weight < 45kg) on 8-28 days, Dexamethasone 5 mg/m2/dose on day 1 and day 8, IT MTX on day 15, 29 (CNS 1, 2 patients), TIT on day 15, 29 (CNS 3 patient)
  Arms: Very high Risk with B-ALL
Drug: Blinatumomab-Salvage 2nd (Very High Risk Group)_4 Weeks — Blinatumomab 28 mcg/day(Weight ≥ 45kg) or 15 mcg/m²/day(Weight < 45kg) on 1-28 days, IT MTX on day 15, 29 (CNS 1, 2 patients), TIT on day 15, 29 (CNS 3 patient)
  Arms: Very high Risk with B-ALL
Drug: Intensification course — <Intensification 1st(3 Weeks)> Etoposide: 100 mg/m2 on day 1, 2, 3, Ifosfamide 3.4 g/m2 on day 1, 2, 3
  <Intensification 2nd(2 Weeks)> Oral 6-mercaptopurine 50 mg/m2/day PO (days 1-14), Methotrexate: 25 mg/m2 on day 1, 8, TIT on day 1
  <Intensification 3rd(3 Weeks)> Ara-C 1.0 g/m2 (days 1-3), Idarubicin: 5mg/m2 (days 1- 3)
  <Intensification 4th(2 Weeks)> Dexamethasone 8 mg/m2/day on days 1-14, Vincristine 2 mg/m2 on days 1 and 8, L-asparaginase 10,000 IU/m2 on days 1 and 8
  Arms: Standard Risk group with B-ALL; Very high Risk with B-ALL
Drug: Maintenance(12 Weeks/Cycle) — Prednisolone: 15 mg/m²/dose(Days 1-5, 29-33, 57-61), Vincristine: 1.5 mg/m²/dose(Day 1, 29, 57), Oral 6-mercaptopurine: 50 mg/m²/dose (Days 1-84), Methotrexate: 20 mg/m²/dose (Days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78), Intrathecal methotrexate (Day 1)
  Arms: Standard Risk group with B-ALL
Procedure: Stem Cell Transplantation — All matters related to hematopoietic stem cell transplantation are subject to each institution's practice.
  Arms: High Risk group with B-ALL; T-ALL

SUMMARY:
This study is open-label, multi-center, prospective study, which targets childhood patients with relapsed acute lymphostatic leukemia including bone marrow recurrence. Aim of this study is to investigate the outcome of NGS MRD based risk stratified treatment for relapsed acute lymphoblastic leukemia in children and adolescents.

DETAILED DESCRIPTION:
The Risk Assessment is classified as follows based on the NGS-MRD results evaluated after EOI(End of Induction).

<Standard Risk>

* Late (Relapse ≥ 1 year after off treatment) B-ALL marrow or Combined relapse AND
* End of induction MRD < 0.01%

<High Risk>

* T-ALL marrow or combined relapse (any timing)
* All other B-ALL marrow or combined relapse cases

<Very High Risk>

• End of Induction BM ≥ M2 AND B -ALL marrow or combined relapse

ELIGIBILITY:
Inclusion Criteria:

* Patients <= 1 year and >22 years of age at the time of relapse will be eligible
* Participants must have a histologic diagnosis of acute lymphoblastic leukemia:

  * B-ALL: Precursor B-cell acute lymphoblastic leukemia
  * T-ALL: Precursor T-cell acute lymphoblastic leukemia
* 1st recurred acute lymphoblastic leukemia patients, recurred parts including marrow. Enrolling patients with combined extra medullary relapse including bone marrow is acceptable. (No limits for extra medullary site) Additionally, subjects whose blast cells in bone marrow are less than 5% (ALL whether type M2 or M3 must be definite)
* Patients who have never received allogeneic stem cell transplant
* Patients who have never received blinatumomab before
* Adequate Renal Function

  -A serum creatinine based on age/gender as follows:

  1 to < 2 years - Male (0.6) Female (0.6) 2 to < 6 years - Male (0.8) Female (0.8) 6 to < 10 years - Male (1) Female (1) 10 to < 13 years - Male (1.2) Female (1.2) 13 to < 16 years - Male (1.5) Female (1.4)

  ≥ 16 years - Male (1.7) Female (1.4)
* Adequate Liver Function defined as a direct bilirubin <3.0 mg/dL
* Adequate Cardiac Function defined as: Shortening fraction of ≥ 27% by echocardiogram, or Ejection fraction of ≥ 50% by echocardiogram
* Lansky (age < 16 years) or Karnofsky (age ≥ 16 years) performance status ≥ 60% at screening
* Patients with a life expectancy of 1 or more year
* Patients who are expected to comply with all required study procedures and follow the study protocol in the opinion of the investigator
* Signed written informed consent and assent forms must be obtained prior to any study procedures

Exclusion Criteria:

* Patients with Burkitt leukemia/lymphoma or mature B-cell leukemia
* Patients with Philadelphia chromosome positive (Ph+) ALL
* Patients with CD19-negative recurrent progenitor B-cell acute lymphoblastic leukemia (non-expression of CD19 in peripheral blood or bone marrow by flow cytometry) are not eligible for administration of Blinatumomab
* In case of relapsed within 1 month after the end of induction with the same 4-drug therapy used in this study
* Patients with mixed phenotype leukemia
* patient who was relapsed within 1 month after the end of induction therapy with the same 4-drug regimen to be used in this study.
* Patients with genetic syndrome: Down syndrome, Bloom syndrome, ataxia-telangiectasia, Fanconi anemia, Kostmann syndrome, Shwachman syndrome bone marrow failure syndrome
* Patients with known HIV
* Female patients who are not proved as infertile or pregnant (Evidence of infertility: History taking of possibilities of pregnancy or urine human chorionic gonadotrophin test negative, amenorrhea more than a year, Natural or artificial (Ex.hormone therapy) menopause status more than a year, surgical sterilization(Ex.Hysterectomy or ovariotomy etc)
* Currently receiving treatment in another investigational drug study or clinical trial
* Evidence of unstable conditions that would pose a risk to subject safety or interfere with the patients' compliance
* Patients with clinically relevant central nervous system (CNS) pathology or active CNS involvement including: unstable epilepsy, uncontrolled seizure, paralysis, aphasia, history of severe brain injury, cerebellar disease, organic brain syndrome, psychosis, coordination/movement disorder
* Known hypersensitivity to drugs or components to be administered: Idarubicin, Etoposide, Ifosfamide, Cytarabine, Vincristine, Mercaptopurine, Blinatumomab

Ages: 1 Year to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2032-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety/Efficacy | through study completion, an average of 9 year
  Patients with relapsed acute lymphoblastic leukemia are being treated after sorted into groups with their potential risk, and disease-free survival rate will be checked.

SECONDARY OUTCOMES:
Disease-free survival rate (Blinatumomab) | through study completion, an average of 9 year
  Blinatumomab is used before transplantation to patients with high-risk group, and then disease-free survival rate will be compared before and after
Disease-free survival rate (standard risk) | through study completion, an average of 9 year
  Patients with standard risk who are not eligible for allogenic stem cell transplantation are given consolidation and maintenance therapies, and disease-free survival rate will compared before and after
Disease-free survival rate (Comparing minimal residual disease) | through study completion, an average of 9 year
  Comparing minimal residual disease negative rate with the study before by adding blinatumomab to patients in high risk group
Death rate related to treatment | through study completion, an average of 9 year
  Children and adolescents who have relapsed acute lymphoblastic leukemia re administered different treatments depending on their assigned groups, and disease-free survival rate will be compared before and after
Death rate related to toxicity | through study completion, an average of 9 year
  Comparing remission rate and occurrence rate of toxicity during re-intervention therapy after changed schedules of idarubicin
Toxicity rate during consolidation therapy | through study completion, an average of 9 year
  Checking occurence rate of toxicity related to treatment during consolidation for patients in low-risk group

CONTACTS AND LOCATIONS:
Overall Officials: Ho Joon Im, Study Chair — Asan Medical Center
Locations (7):
- South Korea (7):
  - Chonnam National University Hwasun Hospital, Hwasun
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul saint Mary's Hospital, Seoul
  - Pusan National University Yangsan Hospital, Yangsan

IPD SHARING:
Plan to Share IPD: No